CLINICAL TRIAL: NCT01286519
Title: Pharmacokinetics of Off Label Pediatric Medications
Status: Recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 10-0865
Record Dates: First submitted 2011-01-21; First posted 2011-01-31 (Estimated); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Off Label Use of Medications in Pediatric Patients
Keywords: pharmacokinetics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The purpose of this study is to measure the level of medicines found in body fluids such as blood, urine, spinal fluid of children.

DETAILED DESCRIPTION:
There is a lack of safety, pharmacokinetic and efficacy data of therapeutic agents in children and infants. Samples used for measurement will be from scavenged samples. i.e. any extra blood/body fluid samples from a test done as part of the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Children less than 8 years of age
* Receiving a therapeutic agent at a dose or for an indication not currently included on the FDA label as part of standard of care

Exclusion Criteria:

* Lack of consent

Ages: 1 Day to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children < 8 years of age currently receiving a therapeutic agent at a dose or for an indication not currently included on the FDA label as part of standard of care
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-07 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) | approximately 10-21 days.The time frame for the outcome measure may vary depending on the length of the course of the medication.
  actual body exposure to drug after a dose of the drug is administered. this is dependent on on the rate of drug elimination divided by plasma concentration of the drug.
Volume of distribution at steady-state | approximately 10-21 days. The time frame for the outcome measure may vary depending on the length of the course of the medication.
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Vss is the apparent volume of distribution at steady-state.
Terminal elimination rate constant (Ke) and Half-Life | approximately 10-21 days. The time frame for the outcome measure may vary depending on the length of the course of the medication.
  Period of time that it takes for the concentration of the drug in the body to be reduced by on-half.
Plasma Clearance | approximately 10-21 days. The time frame for the outcome measure may vary depending on the length of the course of the medication.
  the rate at which the drug is eliminated from the body divided by the plasma concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M. Laughon, MD, MPH, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina NC Children's Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No